CLINICAL TRIAL: NCT06468137
Title: Follow Up of an Online Hearing Support for First-time Hearing Aid Users Using the Swedish I-ACE, Clinical Visit or Nothing
Brief Title: Follow Up of an Online Hearing Support for First-time Hearing Aid Users
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Horselvarden Region Ostergotland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uppföljning
Record Dates: First submitted 2024-04-30; First posted 2024-06-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss; Hearing Impairment; Hearing Disorders
MeSH Terms: conditions — Hearing Loss; Hearing Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Swedish I-ACE (Other): Participants choosing to take part in the Swedish I-ACE as follow-up.
  Interventions: Behavioral: Swedish I-ACE
- Clinical visit (Other): Participants choosing a clinical visit as follow-up.
  Interventions: Behavioral: Clinical visit
- No follow-up (Other): Participants choosing no follow-up.
  Interventions: Other: No follow-up

INTERVENTIONS:
Behavioral: Swedish I-ACE — Rehabilitative programme with focus on communication strategies and problem solving for people with hearing loss.
  Arms: Swedish I-ACE
Behavioral: Clinical visit — Visit in the clinic with focus on audiologic rehabilitation.
  Arms: Clinical visit
Other: No follow-up — Participants choosing no follow-up.
  Arms: No follow-up

SUMMARY:
The main questions the research aims to answer are short- and long-term effects on consequences of hearing loss depending on which type of follow-up the participant chooses.

DETAILED DESCRIPTION:
Investigation of the emotional and social consequences of hearing loss that the participants experience, use of communications strategies, experienced listening in complex sound environments and perceived effectiveness and satisfaction with hearing aids. The goal is also to assess changes in use of communication strategies and the emotional consequences, knowledge and acceptance of hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* People who have participated in NCT06051968 are automatically enrolled to participate in the follow-up according to the study protocol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Hearing Handicap Inventory for the Elderly (HHIE) | Baseline, about 7 weeks post choice of intervention, and 6 months post intervention
  Assessing changes in emotional and social effects of hearing loss, self-perceived activity limitations and participation restrictions. Minimum 0 points to maximum 100 points. Higher score indicates greater emotional and social effects of hearing loss.

SECONDARY OUTCOMES:
The 12-item Speech, Spatial and Qualities of Hearing Scale (SSQ12) | Baseline, about 7 weeks post choice of intervention, and 6 months post intervention
  Assessing experience of listening in complex sound environments. Minimum 0 points to 120 points. Higher score indicates less problems with hearing in the specified situations.
Communication Strategies Scale (CSS) | Baseline, about 7 weeks post choice of intervention, and 6 months post intervention
  Assessing changes in use of verbal, non-verbal and maladaptive communication strategies. Minimum 25 points to maximum 125 points. Higher score indicates a greater use of communication strategies.
The International Outcome Inventory for Hearing Aids (IOI-HA) | Baseline, about 7 weeks post choice of intervention, and 6 months post intervention
  Assessing changes in perceived effectiveness and satisfaction with hearing aids.
  Minimum 7 points to maximum 35 points. Higher score indicates higher perceived effect.
Communication and Acceptance Scale (CAS) | Baseline, about 7 weeks post choice of intervention, and 6 months post intervention
  Assessing changes in use of communication strategies and the emotional consequences, knowledge and acceptance of hearing loss. Minimum 18 points to maximum 90. Higher score indicates a lower impact of the hearing loss.
The International Outcome Inventory for Alternative Interventions (IOI-AI) | Baseline, about 7 weeks post choice of intervention, and 6 months post intervention
  Assessing changes in perceived effectiveness and satisfaction with an alternative intervention, in this case the Swedish I-ACE.
  Minimum 7 points to maximum 35 points. Higher score indicates higher perceived effect.

OTHER OUTCOMES:
Subjective impact of the intervention, reported by the users: Memory of the intervention | Time Frame: 6 months post intervention
  The participants are asked what they remember from their intervention.
Subjective impact of the intervention, reported by the users: Seeking more or other information | Time Frame: 6 months post intervention
  The participants are asked if they searched for more or other information about hearing or hearing aids.
Subjective impact of the intervention, reported by the users: Adverse effects | Time Frame: 6 months post intervention
  The participants are asked if they experienced any adverse effects of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Öberg, Principal Investigator — Horselvarden Region Ostergotland
Locations (1):
- Audiologimottagningen Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No